CLINICAL TRIAL: NCT05283317
Title: The Effect of Mesenchymal Stromal Cells on the Mortality of Patients With Sepsis and Septic Shock: A Promising Therapy
Brief Title: Effect of Mesenchymal Stromal Cells on Sepsis and Septic Shock
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emine ALP MESE, Professor, TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mesenchymal Stromal Cells
Record Dates: First submitted 2022-02-18; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Septic Shock
Keywords: stem cells; sepsis; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients received MSCs (Active Comparator): 10 patients with sepsis and septic shock and received MSCs&standart therapy
  Interventions: Biological: Mesenchymal stem cells
- Patients not received MSCs (No Intervention): 20 patients with sepsis and septic shock and not received MSCs, only received standart therapy

INTERVENTIONS:
Biological: Mesenchymal stem cells — Standard therapy of sepsis as suggested in the guidelines were given to all patients and additionally MSCs treatment was applied to the patients in the study group.
  Arms: Patients received MSCs

SUMMARY:
Methods:Ten patients were enrolled in the study. Adipose derived-MSCs infusions were given (1x 106/ kg, on 1st, 3rd, 5th, 7th and 9th days of therapy) together with Standard therapy. Before the MSCs applications, blood samples were collected for cytokine assessment (TNF-α, IFN-γ, IL-2, IL-4, IL-6, IL-10). The clinical and laboratory improvements were recorded and compared with control groups selected retrospectively.

DETAILED DESCRIPTION:
Study Design and Setting The study was carried out at the Internal Medicine Intensive Care Unit (IMICU) and Anesthesiology and Reanimation Intensive Care Unit (ARICU) at Erciyes University Hospital which is a referral hospital in the Central Anatolia. The study was approved by the Erciyes University Ethics Board (2016/114; Date: 19.02.2016) and Ministry of Health of Turkey. Informed consent from surrogate decision-makers was taken for study participation after confirmation of eligibility criteria.

Patients The study was planned as prospectively. During two years, 10 patients with sepsis and septic shock were included in the study from IMICU and ARICU. Sepsis and septic shock were diagnosed according to the sepsis guidelines [1]. Inclusion criteria for this study were; patients who were between 18-80 years of age and were hospitalized at IMICU and ARICU with the diagnosis of sepsis and septic shock. Exclusion criteria were categorized that patients who were younger than 18-year-old and older than 80 years and were pregnant women or breast-feeding; patients who had terminal stage of cancer, advanced pulmonary disease receiving oxygen at home, advanced pulmonary hypertension (WHO Class III or IV), advanced heart failure (American Heart Association Class III or IV), severe liver disease (Child C), and history of anaphylaxis. Standard therapy of sepsis as suggested in the guidelines [1,2] were given to all patients and additionally MSCs treatment was applied to the patients in the study group. Control patients diagnosed sepsis and septic shock and having similar characteristics for the consideration of severity of disease based on APACHE II score and co-morbid diseases with study group were selected from IMICU and ARICU records retrospectively.

Patients' demographic characteristics, underlying diseases, clinical and laboratory outcomes were recorded.

Source and Application of MSCs MSCs were prepared in Good Manufacturing Practices (GMP) Laboratory of Genome and Stem Cell Center at Erciyes University. Cell production and quality control assessment procedures were carried out according to GMP protocols authorized by the Ministry of Health of Turkey. Allogenic adipose derived MSCs (ADMSCs) which were obtained from a healthy donor were applied to all patients in the study group. Five doses of ADMSCs were applied to the patients at 1st and 3rd day (post-thawed of frozen MSCs cryo-bag), 5th-7th and 9th day (re-plated ADMSCs vials) of therapy. Each dose of ADMSCs was prepared as 1 x 106 ADMSCs/kg. The vials containing ADMSCs were mixed with gentle motions before the usage; thus, it ensured product homogenization. ADMSCs were infused intravenously via central venous line in a physiological saline solution by using a blood transfusion set. The patients were monitored during all these procedures.

Preparation of ADMSCs Sufficient cryo-preserved ADMSCs vials were thawed to provide the required dose for administration. The frozen ADMSCs were thawed and cultured in the Dulbecco's Modified Eagle Medium (DMEM) containing 10% human serum, 1% Penicillin- Streptomycin solution, and 1% stable glutamine (Biological Industries, Kibbutz Beit Haemek, Israel) at 37°C and 5% CO2 incubator which described before [16]. Briefly, ADMSCs were recovered and resuspended in physiological saline solution and transferred to the patient with the temperature-controlled bag. The morphology of cell appearance and the viability were assessed beside the identification of phenotypic characteristics of the cells and microbiological tests. Immunophenotyping characterization of ADMSCs was performed by using flow cytometry analyses (Beckman Coulter, USA) with antibodies against CD45, CD73, CD90, CD105, CD11b, CD19, CD34, CD44 (BD Stem Flow hMSC kit).

Cytokine Analysis Ten ml peripheral venous blood samples were collected before each MSCs infusion at 1st, 3rd,5th, 7thand 9th day of therapy. The serum samples were centrifuged at 5000 rpm for 5 minutes and stored at - 80°C until laboratory analysis. Cytokine level was analyzed with ELISA method by using Human BioSource for (TNF-, IFN- γ, IL-2, IL-4, and IL-10) kits in Robonik Read Well Touch model (Robonik India Pvt Ltd) device.

Clinical and Laboratory Follow-up Clinical findings and laboratory results were recorded at the administration of MSCs infusions at 1st, 3rd, 5th, 7th and 9th days. Patients' demographic characteristics, underlying diseases, clinical and laboratory outcomes were recorded. The patients were monitored for unexpected adverse events. In the clinical follow-up of the patients APACHE II, SOFA (the sequential organ failure assessment score) score, clinical progression and outcome of patients were recorded. As laboratory following, inflammatory markers; C reactive protein (CRP), procalcitonin (PCT) and white blood cell (WBC), bleeding parameters (platelets, INR, fibrinogen), lactate, liver enzymes (AST, ALT), renal functions (creatinine) were also recorded. Laboratory test results were analyzed according to MSCs administration days. The differences of the laboratory tests were compared between the survivor and non-survivor patients according to MSCs therapy days.

Outcomes of the patients were compared with the previous observational study conducted in the same Intensive Care Units (ICUs) as control. The day of death and 0-6th, 7-14th, and 15-28th days were determined as survival status and endpoint. In case of death, the date and cause of death were also recorded.

Statistical Analysis In the study, the results were compared to controls. Statistical analysis was performed using Turcosa software. The relationships between categorical variables were analyzed by chi-square analysis. When parametric assumptions were provided in comparison of numerical variables in two groups, the Student-T test was used and the Mann Whitney U test was in the case that the parametric assumptions did not provide. For the analysis of repeated measurements; Paired Sample T-Test was used for binary comparisons and the Repeated Measures ANOVA test was used for comparison of more than two repeated measurements. The survival probability of the patients during the follow-up period was determined by Kaplan-Maier survival analysis. The effect of age and APACHE II to co-variants analysis were adjusted. p <0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* sepsis and septic shock
* 18-80 years of age

Exclusion Criteria:

* <18-year-old and > 80 years old
* pregnant women or breast-feeding;
* terminal stage of cancer,
* advanced pulmonary disease receiving oxygen at home,
* advanced pulmonary hypertension (WHO Class III or IV),
* advanced heart failure (American Heart Association Class III or IV),
* severe liver disease (Child C),
* history of anaphylaxis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Mortality | 28th days were determined as survival status and endpoint.
  Survival rates of the study group patients were compared with the survival rates of previous observational study conducted in the same Intensive Care Units (ICUs) as control.

SECONDARY OUTCOMES:
Length of stay in the hospital | Through study completion, an average of 1 year
  Length of stay in the hospital of the study patients were compared with length of stay in the hospital previous observational study conducted in the same Intensive Care Units (ICUs) as control.

CONTACTS AND LOCATIONS:
Overall Officials: Emine ALP MESE, Professor, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alp E, Gonen ZB, Gundogan K, Esmaoglu A, Kaynar L, Cetin A, Karakukcu M, Cetin M, Kalin G, Doganay M. The Effect of Mesenchymal Stromal Cells on the Mortality of Patients with Sepsis and Septic Shock: A Promising Therapy. Emerg Med Int. 2022 Jun 24;2022:9222379. doi: 10.1155/2022/9222379. eCollection 2022. PMID 35784641